CLINICAL TRIAL: NCT05908747
Title: Efficacy and Safety of Surufatinib Combined With Gemcitabine and Albumin-bound Paclitaxel in the Peri-operative Treatment of Locally Advanced or Borderline Resectable Pancreatic Cancer: An Exploratory Study
Brief Title: Efficacy and Safety of Surufatinib Combined With Gemcitabine and Albumin-bound Paclitaxel in the Peri-operative Treatment of Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-P105
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — surufatinib; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surufatinib + gemcitabine + nab-paclitaxel (Experimental)
  Interventions: Drug: surufatinib + gemcitabine + nab-paclitaxel

INTERVENTIONS:
Drug: surufatinib + gemcitabine + nab-paclitaxel — surufatinib: 250mg, QD po; nab-paclitaxel: 125mg/m2, I.V., D1/8/15, Q4W; gemcitabine: 1000/m2, ivgtt for more than 30min, D1/8/15, Q4W

SUMMARY:
This study is designed to explore the efficacy and safety of surufatinib combined with gemcitabine and nab-paclitaxel as peri-operative treatment in locally advanced or borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
This is a phase II, multi-centered, open-label study, aims to explore the efficacy and safety of surufatinib (250mg, qd po) combined with gemcitabine (1000mg/m2, I.V, d1/8/15, Q4W) and nab-paclitaxel (125mg/m2, I.V, d1/8/15, Q4W) as peri-operative treatment in locally advanced or borderline resectable pancreatic cancer. Potential therapeutic biomarkers will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high-risk resectable or borderline resectable pancreatic cancer;
* 18-75 years old (including 18 and 75 years old);
* No BRCA1/2 or PALB2 mutation;
* No previous systematic treatment or radiotherapy;
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 6 months;
* At least one measurable lesion according to RECIST version 1.1;
* Adequate organ and bone marrow functions: -Absolute neutrophil count≥1.5x10^9/L; -Platelet count≥100x10^9/L; -Hemoglobin≥9g/dL; -Serum bilirubin≤1.5x the upper limit of normal (ULN); -Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5x ULN; -Serum creatinine≤1.5x ULN or endogenous creatinine clearance rate ≥ 60ml / min; -INR≤1.5×ULN, PT and APTT≤1.5×ULN；
* Women of childbearing age need to take effective contraceptive measures.

Exclusion Criteria:

* With distant metastasis;
* Have received blood transfusion treatment, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF) within 14 days before enrollment;
* Have received any surgery or invasive treatment or operation within 4 weeks before enrollment (except venous catheterization, puncture and drainage, etc.);
* Allergic to the study drug or any of its adjuvants;
* researchers judged clinically significant electrolyte abnormalities;
* History of serious cardiovascular and cerebrovascular diseases: -Cerebrovascular accident (excluding lacunar cerebral infarction, minor cerebral ischemia or transient ischemic attack), myocardial infarction, unstable angina pectoris, and poorly controlled arrhythmia (including QTc interval ≥ 450ms for male and ≥ 470ms for female) occurred within 6 months before the first administration of the study drug (QTc interval was calculated by fridericia formula); -New York Heart Association (NYHA) cardiac function classification > grade II or left ventricular ejection fraction (LVEF) < 50%;
* With active ulcer, intestinal perforation and intestinal obstruction;
* Uncontrollable malignant ascites (defined as ascites that cannot be controlled by diuretics or puncture according to the judgment of the investigator);
* Clinically significant electrolyte abnormalities judged by researchers;
* With active bleeding or obvious evidence of bleeding tendency;
* Hypertension that cannot be controlled by drugs: systolic blood pressure ≥ 150 mmHg and / or diastolic blood pressure ≥ 100 mmHg;
* Women who are pregnant or lactating;
* Urinary protein ≥ ++, or the 24-hour urine protein quantification is greater than 1.0g;
* Concurrent tumors within 5 years (except treated cervical carcinoma in situ, basal cell carcinoma);
* Any disease or state that affects the absorption of drugs, or the subject cannot take oral drugs;
* Known human immunodeficiency virus (HIV) infection;
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×10^4/ml or >2000 IU/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×10^3/m); hepatitis and cirrhosis;
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions that makes the subject not suitable for enrolling according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Surgical complete resection rate (R0) | about 2 years
  This is a complete macroscopic resection of the gross tumor with negative surgical margins

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | about 2 years
  ORR= Complete response rate + partial response rate
Disease Control Rate (DCR) | about 2 years
  DCR= Complete response rate + partial response rate + disease stable rate
Downstaging Rate | about 2 years
  To determine the rate of downstaging after preoperative therapy
Surgical Resection Rate | about 2 years
  To determine the rate of surgical resection after preoperative therapy
Pathological complete response (pCR) rate | about 2 years
  pCR is defined as the absence of residual tumor cells in the pathological examination after resection
Major pathological response (MPR) | about 2 years
  MPR is defined as less than 10% residual tumor after neoadjuvant therapy
Overall survival (OS) | about 5 years
  OS: from the initial date of neoadjuvant therapy to the date of death due to any cause. Patients without documentation of death at the time of analysis will be censored at the last follow-up date. Estimated using Kaplan-Meier method.
Recurrence Free Survival (RFS) | about 3 years
  RFS: from the initial date of neoadjuvant treatment to the first date of radiologic recurrence or death after perioperative treatment.
Disease-free survival (DFS) | about 3 years
  DFS: from the initial date of neoadjuvant treatment to the date of disease recurrence or death, whichever is earlier.
Adverse events (AEs) | about 2 years
  treatment-related adverse events and serious adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Song Gao, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China